CLINICAL TRIAL: NCT04026854
Title: Individual, Organizational and Managerial Determinants of Quality of Life at Work of Psychiatric Nurses and Relief on the Quality of Care
Brief Title: Determinants of the Quality of Work Life of Psychiatric Nurses and Relief on the Quality of Care
Acronym: DETERQVT
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: PHRIP13-PC-DETERQVT
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Quality of Work Life of Psychiatric Nurses; Impact on Quality of Care
Keywords: Quality of life at work;Nurse;Quality of care;psychiatric

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Psychiatric nurses: Nurse with a degree in the state or psychiatric sector. Work in a psychiatric ward that offers full hospitalization, a day hospital (HdJ) or a medico-psychological center (CMP).
  Interventions: Behavioral: Quality of live at work

INTERVENTIONS:
Behavioral: Quality of live at work — The judging criteria will be collected using two questionnaires: a questionnaire sent to the local referent of each center and a questionnaire for each nurse. Because the study is longitudinal (two collections of data), the questionnaires will be completed twice to twelve months apart by the same nurses.

SUMMARY:
Psychological well-being at work is a major public health issue. The number of sick personal leaving hospitals has increased by 10% in five years and the average cost of absenteeism is around 3000 euros per agent per year. These changes are associated with the increase in turnover among nurses, thus raising the question of its impact on the quality of care. Psychological suffering at work is one of the main determinants of intention to leave for nurses.The investigators hypothesize that an improvement in the quality of work life of nurses could lead to greater loyalty, greater motivation of nurses and greater attractiveness within the community. 'institution. Among the publications on psychological well-being at work, few have been interested in the structural aspects of the organization of care and in particular to the variables specific to the caregivers themselves, such as the quality of life at work. Nevertheless, studies carried out in industry show significant and positive links between quality of life at work and performance at work. Thus, it seems appropriate to identify the factors likely to lead to an improvement in the quality of work life of psychiatric nurses and to determine the elements that can help to strengthen it. Moreover, it appears that the field of psychiatry could constitute an ideal field of experimentation. Psychiatry teams treat patients with chronic, severe and debilitating conditions, which are subject to significant social stigmatization, and expose nurses to a high rate of burnout. The organization of psychiatric care is also multidisciplinary. The various care procedures allow caregivers to carry out activities that include more or less significant participation in decision-making. Also, studying the determinants of the quality of working life among psychiatric nurses seems to us an important goal in order to put in place actions to strengthen psychological well-being at work, and thus to reduce turn-over and improve the quality of care.

DETAILED DESCRIPTION:
Psychological well-being at work is a major public health issue. The number of sick personal leaving hospitals has increased by 10% in five years and the average cost of absenteeism is around 3000 euros per agent per year. These changes are associated with the increase in turnover among nurses, thus raising the question of its impact on the quality of care. Psychological suffering at work is one of the main determinants of intention to leave for nurses. The investigators hypothesize that an improvement in the quality of work life of nurses could allow greater loyalty, greater motivation of nurses and greater attractiveness within the institution. Among the publications on psychological well-being at work, few have been interested in the structural aspects of the organization of care and in particular to the variables specific to the caregivers themselves, such as the quality of life at work. Nevertheless, studies carried out in industry show significant and positive links between quality of life at work and performance at work. Thus, it seems appropriate to identify the factors likely to lead to an improvement in the quality of life at work of psychiatric nurses and to determine the elements that can help reinforce it. Moreover, it appears that the field of psychiatry could constitute an ideal field of experimentation. Psychiatry teams treat patients with chronic, severe and disabling conditions, which are subject to significant social stigma, and expose nurses to a high rate of burnout. The organization of psychiatric care is also multidisciplinary. The various care procedures allow caregivers to carry out activities that include more or less significant participation in decision-making. Also, studying the determinants of the quality of life at work among psychiatric nurses seems to be an important goal in order to implement actions to strengthen psychological well-being at work, and thus reduce turnover and to improve the quality of care.

The main objective is to identify the individual, organizational and managerial factors that can explain changes in the quality of work life of psychiatric nurses.

To study the link between changes in the quality of work life of nurses and the quality of care delivered to patients.

Study the effects of a change in the quality of work life of nurses on turnover.

ELIGIBILITY:
Inclusion Criteria:

* Nurse with a degree in the state or psychiatric sector.
* Working in a psychiatric ward that offers full hospitalization, a day hospital (HdJ) or a medico-psychological center (CMP).

Exclusion Criteria:

* N/A

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Nurse with a degree in the state or psychiatric sector.
  * Working in a psychiatric ward that offers full hospitalization, a day hospital (HdJ) or a medico-psychological center (CMP).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Measuring the quality of work life of nurses by the French version of the quality of life (QOL) at work scale of Elizur and Shye (1990). | 1 year
  The quality of work life of nurses as measured by the French version of the quality of life at work scale of Elizur and Shye (1990). This scale assesses four dimensions of quality of life at work. It has 16 items that can be answered using a Likert scale ranging from 1 (very little) to 6 (mostly). The higher the score, the better the quality of life at work.

SECONDARY OUTCOMES:
Measuring psychological well-being at work using the scale of Gilbert, Dagenais-Desmarais and Savoie (2011). | 1 year
  Psychological well-being at work measure using the scale of Gilbert, Dagenais-Desmarais and Savoie (2011).This scale assesses psychological well-being at work. It has 22 items that can be answered using a Likert scale ranging from 1 (never) to 5 (almost always). The higher the score, the better the quality of life at work.
Measuring job satisfaction using an adaptation of the job satisfaction scale of Fouquereau and Rioux (2002). | 1 year
  Job satisfaction measure using an adaptation of the job satisfaction scale of Fouquereau and Rioux (2002).It has 5 items that can be answered using a Likert scale ranging from 1 (very unsatisfied) to 5 (very satisfied). The higher the score, the better the quality of life at work.
Measuring work engagement using the French version of UWES-9 (Schaufeli, Bakker, Salanova, 2006). | 1 year
  Work engagement measured using the French version of Utrecht Work Engagement Scale (UWES-9) (Schaufeli, Bakker, Salanova, 2006).It has 9 items that can be answered using a Likert scale ranging from 1 (never) to 6 (always). The higher the score, the better the work engagement.
Measuring the satisfaction of psychological needs at work using the satisfaction scale of the psychological needs of Gillet, Rosnet and Vallerand (2008). | 1 year
  The satisfaction of psychological needs at work measured using the satisfaction scale of the psychological needs of Gillet, Rosnet and Vallerand (2008).It has 28 items that can be answered using a Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). The higher the score, the better the satisfaction.
Measuring the feeling of self-efficacy from the questionnaire referring to specific behaviors in General Self-Efficacy Scale (GSE) Nagels (2008) | 1 year
  The feeling of self-efficacy (GSE) measured from the questionnaire referring to specific behaviors in Nagels (2008); It has 10 items that can be answered using a Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree). The range is from 10 to 40 points. The higher the score, the better feeling of self-efficacy.
Measuring thetransformational leadership using the Global Transformational Leasership scale (GTL) developed by Carless, Wearing and Mann (2000). | 1 year
  Transformational leadership measured using the GTL scale developed by Carless, Wearing and Mann (2000). It has 7 items that can be answered using a Likert scale ranging from 1 (not at all) to 5 (frequently, if not always). The higher the score, the better the Transformational leadership
Measuring the support for autonomy using a version adapted to the work context of the Measuring the Perceived Autonomy Support Scale for Exercise Settings (PASSES) of Gillet, Vallerand, Paty, Gobancé and Berjot (2010). | 1 year
  Support for autonomy measured using a version adapted to the work context of the PASSES scale; Gillet, Vallerand, Paty, Gobancé and Berjot (2010).It has 12 items that can be answered using a Likert scale ranging from 1 (strongly disagree)) to 7 (strongly agree).The higher the score, the better the perceived autonomy.
Measuring the personality using Big Five Inventory (BFI) by John, Donahue and Kentle (1991). | 1 year
  Personality measured using BFI by John, Donahue and Kentle (1991).It has 44 items that can be answered using a Likert scale ranging from 1 (disagree a lot) to 5 (agree a lot). The higher the score, the better the personality
Measuring the well-treatment by a self-evaluation of patient well-being practices, Terrien,Anthoine and Mouret (2012). | 1 year
  Well-treatment measured by a self-evaluation of patient well-being practices, Terrien, Anthoine and Mouret (2012).
  It has 16 items that can be answered using a Likert scale ranging from 1 (always) to 5 (never ). The lower the score, the better the well-treatement.
  .

CONTACTS AND LOCATIONS:
Overall Officials: Pierre CHEYROUX, Study Director — University Hospital of TOURS